CLINICAL TRIAL: NCT01633684
Title: Type 1 DM Effect on BMD: a Longitudinal Study in Adults
Brief Title: Type 1 Diabetes Mellitus Effect on Bone Mineral Density
Status: Completed | Type: Observational
Sponsor: Creighton University (Other)
Responsible Party: Sponsor
Other Study IDs: Creighton 14
Record Dates: First submitted 2012-07-02; First posted 2012-07-04 (Estimated); Last update posted 2014-10-31 (Estimated); Status verified 2014-10

CONDITIONS: Diabetes Mellitus; Osteoporosis
Keywords: diabetes mellitus; bone
MeSH Terms: conditions — Diabetes Mellitus; Osteoporosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — We will be storing serum samples. No genetic tests will be performed on these.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Diabetes: patients with Type 1 Diabetes Mellitus
- Control: Age and sex matched control subjects

SUMMARY:
Because the diabetics are fracturing at a younger age than the general population (12), this leads us to believe there are significant factors that lead to fracture in Type 1 diabetes mellitus (DM) other than bone mineral density (BMD). Very little longitudinal data exists on BMD in adults with Type 1 DM and the effects of glucose control on BMD. No longitudinal data exists on pQCT in adults with Type 1 DM.

Hypothesis: Adult subjects with diabetes and poor glucose control will lose bone mineral density (BMD) as measured by DXA compared to age and sex matched healthy controls.

DETAILED DESCRIPTION:
Because the diabetics are fracturing at a younger age than the general population(12), this leads us to believe there are significant factors that lead to fracture in Type 1 DM other than BMD. Very little longitudinal data exists on BMD in adults with Type 1 DM and the effects of glucose control on BMD. No longitudinal data exists on pQCT in adults with Type 1 DM.

Hypothesis: Adult subjects with diabetes and poor glucose control will lose bone mineral density (BMD) as measured by DXA compared to age and sex matched healthy controls.

ELIGIBILITY:
Inclusion Criteria:

* diabetic patients must have completed Visit 1 of the previous study.

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Subjects who have Type 1 DM and their age and sex matched control and have been enrolled in a study of Type 1 DM and bone and had a baseline DXA and pQCT during the last 4 years. Persons that completed visit 1 for the previous study and had a DXA and pQCT done will be invited back for repeat DXA and pQCT measurement. If a diabetic patient does not have an age and sex matched control or their control does not want to be in the longitudinal study a new age and sex matched control will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 123 (Actual)
Dates: Start 2012-08; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Bone mineral Density | 5 years
  Bone mineral density will be measured yearly for 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Laura Armas, MD,MS, Principal Investigator — Creighton University
Locations (1):
- Creighton University, Omaha, Nebraska, United States